CLINICAL TRIAL: NCT03724370
Title: Using Telehealth to Improve Outcomes in Veterans at Risk for Suicide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, Gretchen L. Haas, PhD, PI, VA Pittsburgh Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LSRG-0-060-15
Record Dates: First submitted 2018-08-28; First posted 2018-10-30 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TES+ VHA-SRM (Experimental): Telehealth monitoring system (TES) will be added to the VA suicide risk management system (VHA-SRM)
  Interventions: Behavioral: Telehealth Monitoring System; Other: VHA-SRM
- VHA-SRM (Active Comparator): VHA-SRM will be active comparator
  Interventions: Other: VHA-SRM

INTERVENTIONS:
Behavioral: Telehealth Monitoring System — TES will be conducted daily via Interactive Voice Response System (IVRS) during the 12 week study period.TES will be added to VHA-SRM.
  Arms: TES+ VHA-SRM
Other: VHA-SRM — Veterans Health Administration Suicide Risk Management supportive services will be provided to participant during the 12 weeks of study participation.

SUMMARY:
Overview. The investigators will randomize 120 Veterans in this 3-site trial over 16 months. Eligible Veterans will include those to be discharged for a hospitalization for suicidal ideation. Baseline data collection and randomization will occur at discharge. The 3 month intervention will have study assessments at 2, 4, 8, and 12 weeks post-discharge. The study's primary outcome measure is suicidal ideation (measured with the Beck Scale for Suicidal Ideation[BSS] and secondarily with the Columbia Scale for Suicidality C-SSRS).

Intervention Components. The control condition will consist of Veterans randomized to VHA-SRM (Suicide Risk Monitoring). The experimental condition will be the telehealth system (TES) + VHA-SRM (Suicide Risk Monitoring) intervention. Veterans randomized to the telehealth system will receive the Interactive Voice Response (IVR) system monitoring in addition to VHA-SRM and will receive training on how to use the TES from the research coordinator. Veterans can access the IVR as a telephonic device accessed by a local or toll-free number and can use a 'plain old telephone system' (POTS), Cellular phone or Internet phone connected to their phone service provider. Participants will be instructed to interact daily with the TES system daily. Because of safety concerns, questions pertaining to suicidal behavior will be asked daily; to avoid repetition, all other questions will be asked every 3rd day. Once participants complete the questions on the telehealth device, their responses will be automatically uploaded and checked by trained VA Pittsburgh Healthcare System (VAPHS) nurses every 4 hours, during regular daytime hours of 9-5. VAPHS will serve as the central site retrieving downloads for all sites. Color-coded risk triage level designations based on potential responses, provide guidance regarding next steps. The protocol for assessing suicidal patients will follow standard VA procedures, outlined in each medical center's safety plan for suicidal patients.

DETAILED DESCRIPTION:
A subject will be considered enrolled after they sign the consent form, but prior to the initiation of study procedures. After enrollment, subjects will undergo baseline assessments and will be randomized prior to discharge from index hospitalization. The study aims to randomize 120 Veterans in 3-sites over 16-20 months.

Once a Veteran has been identified and referred, a member of the study team will meet with the Veteran on the inpatient unit to obtain consent. The baseline visit may take place all at once or on different days while patients are on the inpatient service. The investigators will attempt to perform baseline assessments as close to discharge as possible in order to obtain a true baseline assessment. However, the investigators may not be able to be certain regarding time of discharge and if this is the case or if discharge is extended, the baseline will be repeated one or more times to ensure that we have baseline data close to the time of discharge.

To assess eligibility, the following will be administered:

1. Folstein Mini Mental Status Exam to assess cognitive impairment.
2. The Beck Scale for Suicidal Ideation (SSI) to assess suicidal ideation.
3. The 17 item Hamilton Depression Rating Scale (HAM-17) to rate depressive symptoms.
4. The Mini International Neuropsychiatric Interview (MINI) to determine diagnoses.

Also administered will be the Sociodemographics Form, Columbia Scale for Suicidality (C-SSRS), Beck Hopelessness Scale©, Brief Addiction Monitor (BAM), Brief Emotional Closeness Questionnaire (ECQ), Brief Medication Questionnaire (BMQ), Hamilton Depression Rating Scale (HAM-D17), Clinical Global Impressions (CGI), and the Medical Outcomes Studies Social Support Survey (MOS-36). Participants that have a diagnosis of Schizophrenia(SZ) or Schizoaffective(SZA) disorder will additionally receive the Scales for the Assessment of Positive and Negative Symptoms (SAPS and SANS). These may be completed any time during the inpatient hospitalization.

In order to obtain a true baseline, these assessments may be administered more than once to obtain the measure as close to the participant's discharge as possible.

Eligible Veterans who complete the assessments will be randomized close to the time of discharge in blocks and stratified by site. When a participant is ready to be randomized, a non-blinded study staff member will access the randomization scheme database/spreadsheet. Staff will click a button to "randomize" and to determine which group they are in. The slot with the group will be provided to the staff member and documented in the database/spreadsheet with the subject identifier (ID) and the date of randomization. At least one of the assessors will be masked, or "blinded," to treatment. The control condition will consist of Veterans randomized to VHA suicide risk management (VHA-SRM). The experimental condition will be the telehealth + VHA suicide risk management (TES+VHA-SRM) intervention.

The intervention is an Interactive Voice Response system, provided by vendor AMC Health. See Appendices 3 and 4. Using the scripts in the protocol, the system will call the patient at the time of day requested by the patient, and ask the questions on the schizophrenia script(for Veterans with schizophrenia or schizoaffective disorder) or the questions on the depression script for all other patients. The patient will answer each question numerically, by either pressing a number or stating the number to the system. The responses will be accessed through a secure web portal maintained by AMC Health, and reviewed Q4 hours by the VAPHS nurses.

The study team will aim to keep an assessor blinded to treatment. This assessor will administer the assessments over follow up.

Veterans randomized to TES+VHA-SRM will receive the IVR system in addition to VHA-SRM and will receive training on how to use the TES from non-blinded research staff, including instructions to contact their providers for any clinical concerns, as well as the research team, or the Veterans Crisis Line. Veterans can use IVR as telephonic device accessed by a local or toll-free number and can use a Plain Old Telephone System (POTS) device connected to their landline or Cellular phone or Internet Protocol phone connected to their phone service provider. Participants will be instructed to interact daily with the TES system daily. Patients will receive the dialogue specific for depression unless they have a diagnosis of SZ/SZA, in which case they will receive the SZ/SZA dialogue. Because of safety concerns, questions pertaining to suicidal behavior will be asked daily; to avoid repetition, all other questions will be asked every 3rd day. Once participants complete the questions on the telehealth device, their responses will be automatically uploaded and checked by trained VAPHS nurses every 4 hours, during regular daytime work hours, 9-5. VAPHS will serve as the central site retrieving downloads for all sites. The website will include responses with color-coded risk triage level designations and staff will receive guidance regarding next steps based on these color codes. The protocol for assessing suicidal patients will follow standard VA procedures, outlined in each medical center's safety plan for suicidal patients.

Veterans randomized to TES+VHA-SRM will be asked to use the IVR system once within a 24 hour period. If an IVR session is not completed within this time frame, the system will automatically call the participant the next morning at a phone number provided by the participant. If the IVR session is not successfully completed after the automatic session is sent, the VAPHS nursing staff will be alerted to this at 12 pm, noon on the website. They will contact the participant's clinician or study staff at that particular site to alert them they have not completed an IVR session. Study staff will track adherence rates to the IVR system.

Veterans randomized to TES+VHA-SRM will have adherence to the telehealth system tracked daily. All subjects will have appointment adherence tracked for 12 weeks post discharge from index hospitalization and psychiatric hospitalizations will be tracked for 12 months post-randomization.

The study team may call the patient's psychiatrist, other clinician, or a significant other (i.e. a family member), or another significant other in the community who the subject has identified and has provided consent for the study team to contact. The team will only contact someone other than the subject's psychiatrist or other clinician if the team has not been able to reach the subject for 48 hours.

All subjects will come in at weeks 2, 4, 8 and 12 following discharge either at the VAPHS outpatient clinics, the VA community based outpatient clinics, Vet centers. They may come in within a 2-week window before or after the expected assessment date.

The following assessments will be administered at follow up: SSI, CSS, HAM-D17, Beck Hopeless Scale, National Institute of Drug Abuse (NIDA) Brief Substance Use Questionnaire, BMQ, and CGI. Participants that have a diagnosis of Schizophrenia or Schizoaffective disorder will additionally receive SAPS and SANS.

In addition to the assessments listed above, week 12 will also administer MOS-36 for all participants and the After Scenario questionnaire for those randomized to TES+VHA-SRM.

During the course of the study, appointment adherence will be tracked for the 12 week of active participation and psychiatric hospitalizations will be tracked for 12 months post-randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans > 18 years old;
2. any diagnosis as long as participants exhibit at least mild depressive symptoms, i.e., a Hamilton 17-item depression 30 score >8; this includes patients with schizophrenia/schizoaffective disorder;
3. score >1 on items 4 or 5 on the SSI ; which assesses active or passive suicidal ideation, respectively.-

Exclusion Criteria:

1. Cognitive problems that would interfere with Veterans' ability to manage the TES system (e.g., neurocognitive d/o, significant traumatic brain injury, or a Folstein Mini Mental Status Exam score <22) or serious motor dexterity problems;
2. Veterans without phone access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-12-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Scale for Suicidal Ideation (BSS). Aaron T. Beck, copyright 1991. | At every visit: screen, baseline(s), week 2,4,6,8,12; timeframe is the past week, including today.
  Continuous scale assessing suicidal ideation. Scores will range from 0 to 42, with lower scores indicating less suicidal ideation.

SECONDARY OUTCOMES:
Change in Columbia Suicide Severity Rating Scale (C-SSRS). Posner, K; Brent, D; Lucas, c; Gould, M; Stanley, B; Brown, G; Fisher, P; Zelazny, J; Burke, A; Oquendo, M; Mann, J. | At every visit: screen, baseline(s), week 2,4,6,8,12; time frame includes lifetime and since last visit.
  Scale assessing suicidal ideation, attempts and behaviors. Mean change in suicidal behavior minimum total score 0, maximum total score 5, higher total scores indicate more suicidal behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen L Haas, Ph.D., Principal Investigator — VA Pittsburgh Healthcare System
Locations (2):
- United States (2):
  - VA NY Harbor Healthcare System, Manhattan Campus, New York, New York
  - James J. Peters Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kemp, J & Bossarte R. (2013). Suicide data report: 2012. Department of Veterans Affairs, Mental Health Services, Suicide Prevention Program.
- [Background] Bruce ML. Suicide risk and prevention in veteran populations. Ann N Y Acad Sci. 2010 Oct;1208:98-103. doi: 10.1111/j.1749-6632.2010.05697.x. PMID 20955331
- [Background] Zivin K, Kim HM, McCarthy JF, Austin KL, Hoggatt KJ, Walters H, Valenstein M. Suicide mortality among individuals receiving treatment for depression in the Veterans Affairs health system: associations with patient and treatment setting characteristics. Am J Public Health. 2007 Dec;97(12):2193-8. doi: 10.2105/AJPH.2007.115477. Epub 2007 Oct 30. PMID 17971541
- [Background] Report of the Blue Ribbon Work Group on Suicide Prevention in the Veteran Population. Washington, DC: U.S. Department of Veterans Affairs.
- [Background] Department of Veterans Affairs, Inpatient Mental Health Services, VHA Handbook 1160.06, 9/16/2013
- [Background] Desai RA, Dausey DJ, Rosenheck RA. Mental health service delivery and suicide risk: the role of individual patient and facility factors. Am J Psychiatry. 2005 Feb;162(2):311-8. doi: 10.1176/appi.ajp.162.2.311. PMID 15677596
- [Background] Valenstein M, Eisenberg D, McCarthy JF, Austin KL, Ganoczy D, Kim HM, Zivin K, Piette JD, Olfson M, Blow FC. Service implications of providing intensive monitoring during high-risk periods for suicide among VA patients with depression. Psychiatr Serv. 2009 Apr;60(4):439-44. doi: 10.1176/ps.2009.60.4.439. PMID 19339317
- [Background] Hoffmire CA, Kemp JE, Bossarte RM. Changes in Suicide Mortality for Veterans and Nonveterans by Gender and History of VHA Service Use, 2000-2010. Psychiatr Serv. 2015 Sep;66(9):959-65. doi: 10.1176/appi.ps.201400031. Epub 2015 May 1. PMID 25930036
- [Background] The Assessment and Management of Risk for Suicide Working Group. 2013. VA/DoD Clinical Practice Guideline for Assessment and Management of Patients at Risk for Suicide. Retrieved from: http://www.healthquality.va.
- [Background] Blow FC, Bohnert AS, Ilgen MA, Ignacio R, McCarthy JF, Valenstein MM, Knox KL. Suicide mortality among patients treated by the Veterans Health Administration from 2000 to 2007. Am J Public Health. 2012 Mar;102 Suppl 1(Suppl 1):S98-104. doi: 10.2105/AJPH.2011.300441. PMID 22390612
- [Background] McCarthy JF, Valenstein M, Kim HM, Ilgen M, Zivin K, Blow FC. Suicide mortality among patients receiving care in the veterans health administration health system. Am J Epidemiol. 2009 Apr 15;169(8):1033-8. doi: 10.1093/aje/kwp010. Epub 2009 Feb 27. PMID 19251753
- [Background] Gibbons RD, Brown CH, Hur K, Davis J, Mann JJ. Suicidal thoughts and behavior with antidepressant treatment: reanalysis of the randomized placebo-controlled studies of fluoxetine and venlafaxine. Arch Gen Psychiatry. 2012 Jun;69(6):580-7. doi: 10.1001/archgenpsychiatry.2011.2048. PMID 22309973
- [Background] Almeida OP, Pirkis J, Kerse N, Sim M, Flicker L, Snowdon J, Draper B, Byrne G, Goldney R, Lautenschlager NT, Stocks N, Alfonso H, Pfaff JJ. A randomized trial to reduce the prevalence of depression and self-harm behavior in older primary care patients. Ann Fam Med. 2012 Jul-Aug;10(4):347-56. doi: 10.1370/afm.1368. PMID 22778123
- [Background] Tarrier N, Taylor K, Gooding P. Cognitive-behavioral interventions to reduce suicide behavior: a systematic review and meta-analysis. Behav Modif. 2008 Jan;32(1):77-108. doi: 10.1177/0145445507304728. PMID 18096973
- [Background] Valenstein M, Kim HM, Ganoczy D, Eisenberg D, Pfeiffer PN, Downing K, Hoggatt K, Ilgen M, Austin KL, Zivin K, Blow FC, McCarthy JF. Antidepressant agents and suicide death among US Department of Veterans Affairs patients in depression treatment. J Clin Psychopharmacol. 2012 Jun;32(3):346-53. doi: 10.1097/JCP.0b013e3182539f11. PMID 22544011
- [Background] Bostwick JM, Pankratz VS. Affective disorders and suicide risk: a reexamination. Am J Psychiatry. 2000 Dec;157(12):1925-32. doi: 10.1176/appi.ajp.157.12.1925. PMID 11097952
- [Background] Godleski L, Nieves JE, Darkins A, Lehmann L. VA telemental health: suicide assessment. Behav Sci Law. 2008;26(3):271-86. doi: 10.1002/bsl.811. PMID 18548515
- [Background] Valenstein M, Kim HM, Ganoczy D, McCarthy JF, Zivin K, Austin KL, Hoggatt K, Eisenberg D, Piette JD, Blow FC, Olfson M. Higher-risk periods for suicide among VA patients receiving depression treatment: prioritizing suicide prevention efforts. J Affect Disord. 2009 Jan;112(1-3):50-8. doi: 10.1016/j.jad.2008.08.020. Epub 2008 Oct 22. PMID 18945495
- [Background] While D, Bickley H, Roscoe A, Windfuhr K, Rahman S, Shaw J, Appleby L, Kapur N. Implementation of mental health service recommendations in England and Wales and suicide rates, 1997-2006: a cross-sectional and before-and-after observational study. Lancet. 2012 Mar 17;379(9820):1005-12. doi: 10.1016/S0140-6736(11)61712-1. Epub 2012 Feb 2. PMID 22305767
- [Background] Mishara BL, Chagnon F, Daigle M, Balan B, Raymond S, Marcoux I, Bardon C, Campbell JK, Berman A. Which helper behaviors and intervention styles are related to better short-term outcomes in telephone crisis intervention? Results from a Silent Monitoring Study of Calls to the U.S. 1-800-SUICIDE Network. Suicide Life Threat Behav. 2007 Jun;37(3):308-21. doi: 10.1521/suli.2007.37.3.308. PMID 17579543
- [Background] Kasckow J, Zickmund S, Rotondi A, Mrkva A, Gurklis J, Chinman M, Fox L, Loganathan M, Hanusa B, Haas G. Development of telehealth dialogues for monitoring suicidal patients with schizophrenia: consumer feedback. Community Ment Health J. 2014 Apr;50(3):339-42. doi: 10.1007/s10597-012-9589-8. Epub 2013 Jan 10. PMID 23306676
- [Background] De Vito Dabbs A, Myers BA, Mc Curry KR, Dunbar-Jacob J, Hawkins RP, Begey A, Dew MA. User-centered design and interactive health technologies for patients. Comput Inform Nurs. 2009 May-Jun;27(3):175-83. doi: 10.1097/NCN.0b013e31819f7c7c. PMID 19411947
- [Background] Rubin J. (1994). Handbook of Usability Testing: How to Plan, Design, and Conduct Effective Tests. New York, NY: John Wiley & Sons, Inc.
- [Background] Gould JD, Lewis C. (1985). Designing for usability: key principles and what designers think. Commun ACM. 2:300-311.
- [Background] Kasckow J, Zickmund S, Rotondi A, Welch A, Gurklis J, Chinman M, Fox L, Haas GL. Optimizing Scripted Dialogues for an e-Health Intervention for Suicidal Veterans with Major Depression. Community Ment Health J. 2015 Jul;51(5):509-12. doi: 10.1007/s10597-014-9775-y. Epub 2014 Oct 24. PMID 25342076
- [Background] Kasckow J, Gao S, Hanusa B, Rotondi A, Chinman M, Zickmund S, Gurklis J, Fox L, Cornelius J, Richmond I, Haas GL. Telehealth Monitoring of Patients with Schizophrenia and Suicidal Ideation. Suicide Life Threat Behav. 2015 Oct;45(5):600-611. doi: 10.1111/sltb.12154. Epub 2015 Feb 17. PMID 25688921
- [Background] Beck AT, Kovacs M, Weissman A. Assessment of suicidal intention: the Scale for Suicide Ideation. J Consult Clin Psychol. 1979 Apr;47(2):343-52. doi: 10.1037//0022-006x.47.2.343. No abstract available. PMID 469082
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Beck AT, Weissman A, Lester D, Trexler L. The measurement of pessimism: the hopelessness scale. J Consult Clin Psychol. 1974 Dec;42(6):861-5. doi: 10.1037/h0037562. No abstract available. PMID 4436473
- [Background] MacArthur Sociodemographic Questionnaire. (2008). The Regents of the University of California
- [Background] Screening for Drug Use in General Medicine: Resource Guide. National Institute on Drug Abuse.
- [Background] Andreason N. Scale for Assessment of Positive Symptoms (SAPS). (1984). University of Iowa, Department of Psychiatry, Iowa City, Iowa.
- [Background] Svarstad BL, Chewning BA, Sleath BL, Claesson C. The Brief Medication Questionnaire: a tool for screening patient adherence and barriers to adherence. Patient Educ Couns. 1999 Jun;37(2):113-24. doi: 10.1016/s0738-3991(98)00107-4. PMID 14528539
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] American Psychiatric Association. Structured Clinical Interview for DSM-5 (SCID-5). Arlington, 2015.